CLINICAL TRIAL: NCT00266058
Title: Pharmacokinetic Interactions Between Antiretroviral Agents, Lopinavir/Ritonavir and Efavirenz and Antimalarial Drug Combination, Artemether/Lumefantrine
Brief Title: Drug Interaction Study Between Antimalarial and Anti-HIV Medications
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Fran Aweeka, Prinicpal Investigator, University of California, San Francisco
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: AAKE99
Record Dates: First submitted 2005-12-14; First posted 2005-12-15 (Estimated); Last update posted 2013-06-06 (Estimated); Status verified 2013-05

CONDITIONS: HIV Infections; Malaria
Keywords: healthy; controls; research; clinical; study; pharmacokinetic; PK; HIV; malaria
MeSH Terms: conditions — HIV Infections; Malaria | interventions — Lopinavir; Ritonavir; efavirenz; Artemether, Lumefantrine Drug Combination

ARMS (2):
- Lopinavir/ritonavir, artemethr/lumefantrine (Active Comparator): Determination of the antimalarial drug levels artemether/lumefantrine in the absence and in the presence of co-administered antiretrovirals lopinavir and ritonavir.
  Interventions: Drug: Lopinavir/Ritonavir, Efavirenz, Artemether/lumefantrine
- efavirenz, artemether, lumefantrine (Active Comparator): Determination of the antimalarial drug levels artemether/lumefantrine in the absence and in the presence of co-administered antiretroviral efavirenz.
  Interventions: Drug: Lopinavir/Ritonavir, Efavirenz, Artemether/lumefantrine

INTERVENTIONS:
Drug: Lopinavir/Ritonavir, Efavirenz, Artemether/lumefantrine — participants receive a total of 6 doses of artemether(80mg)/lumefantrine(480mg)for baseline PK evaluation. This is followed by a 26-day course of either efavirenz(600mg) once daily or lopinavir/ritonavir (400mg/100mg) twice daily and additional 6 doses of artemether/lumefantrine to determine the pharmacokinetics of the antimalarial medications in the context of antiretrovirals. The participants undergo at least a 14 day washout period (between the last baseline PK blood draw and the initiation of antiretrovirals)

SUMMARY:
The purpose of this study is to find out whether taking certain anti-HIV medicines with certain antimalarial medicines affects the amount of the medicines in the blood.

The study medicines that will be used are artemether/lumefantrine (antimalarial medication) and lopinavir/ritonavir or efavirenz (anti-HIV medications). Artemether/lumefantrine is not approved by the United States Food and Drug Administration (FDA) but is recommended as standard of care medical treatment for malaria in Africa and Asia. Lopinavir/ritonavir and efavirenz are approved by the FDA. Artemether/lumefantrine and lopinavir/ritonavir or efavirenz may need to be used together to treat children in Africa and Asia. We seek to learn about whether or not the use of these medicines together results in a change in blood levels of any of these medicines. The information obtained from this study will help doctors to provide a better treatment to children and adults with malaria and HIV.

DETAILED DESCRIPTION:
The study involves 5 non-consecutive overnight stays and 14 additional outpatient visits at the San Francisco General Hospital Research Center.

ELIGIBILITY:
Inclusion Criteria:

* Absence of HIV infection prior to study entry
* Within 20% (+/-) of ideal body weight and must weigh at least 50kg
* Healthy subjects without evidence of acute or chronic illnesses, including diabetes, high blood pressure, coronary artery disease, psychiatric illnesses, liver or kidney impairment

Exclusion Criteria:

* Use of illicit drugs or alcohol that could interfere with the completion of the study.
* Use of any over- the- counter or prescribed drugs unless approved by the principal investigator or study physician.
* Pregnant or breast- feeding.
* History of acute or chronic illnesses, such as diabetes, high blood pressure, coronary artery disease, psychiatric illnesses, liver or kidney impairment.
* Evidence of acute illness.
* Family history of congenital prolongation of QTc interval or with any conditions known to prolong QTc interval, such as cardiac arrhythmias, bradycardia or severe heart disease
* History of electrolyte abnormalities.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2005-12; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic assessment of potential drug-drug interactions of antimalarials and antiretroviral agents. | Intensive serial PK sampling of antimalarials conducted on study day 4 (without antiretrovirals) and study day 31 (in the context of antiretrovirals

CONTACTS AND LOCATIONS:
Overall Officials: Francesca Aweeka, Pharm.D., Principal Investigator — University of California, San Francisco
Locations (1):
- San Francisco General Hospital, San Francisco, California, United States